CLINICAL TRIAL: NCT00817960
Title: Effects of Methylphenidate on Postural Stability of Old Adults Under Single and Dual Task Conditions.
Brief Title: Effects of Ritalin on Postural Stability of Old Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SOR476508CTIL; MZ4765
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2008-12

CONDITIONS: Postural Imbalance
Keywords: Dual tasking; Postural Control; Methylphenidate (Ritalin); old adults
MeSH Terms: interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Methylphenidate (Experimental)
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate — The effect of ritalin on postural stability of old adults (65 years old and over) will be measured using RCT study design

SUMMARY:
Experimental design overview The proposed project is a prospective experimental study design. independent old adults(age 65 years old and older) who do not suffer from balance problems willing to participate in the study will be tested with well-established measuring techniques of Balance control before and 2 hours after taking of Methylphenidate (Ritalin) in the movement and Rehabilitation Laboratory at BGU. An automated algorithm will be used to extract standardized stabilogram-diffusion parameters from each of the COP data sets collected during quiet standing. These parameters include diffusion coefficients, critical displacement, critical time and scaling exponents for both lateral and anterior-posterior sway directions (Collins & De Luca, 1993). For each of the conditions (before and 1 hour after the use of Ritalin) in three task conditions single task; dual task (concentrating and identifying specific music); and just Listening to a relaxing music. Participants will be required to stand on the platform 10 times for 30 s. For each trial, they will be instructed to sway as little as possible.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years old and older
* independent elderly adults
* do not suffer from balance prblems
* minimental score 24 and above

Exclusion Criteria:

* old adults who suffer from neurological disease or stroke
* old adults who suffer from psychiatric state
* old adults who suffer from orthopedic condition (1/2 a year after a fracture in the lower limb)
* old adults who suffer from heart conditions
* old adults who suffer from blindness

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Postural sway measures | Time 1: pre test' and hour later time 2: post testinng proceedure

CONTACTS AND LOCATIONS:
Overall Officials: Itshak Melzer, PhD, Principal Investigator — Ben-gurion University of the Negev, Beer-Sheva, Israel; Zmir Shorer, m, Study Chair — Soroka University Medical Centar; Yan Press, MD, Study Director — Soroka University Medical Center
Locations (1):
- SorokaUMC, Beersheba, Israel, Israel